CLINICAL TRIAL: NCT04544514
Title: Earliest Lung Ultrasound Time for Predicting the Need of Surfactant
Status: Completed | Type: Observational
Sponsor: Gozdem Kayki (Other)
Responsible Party: Sponsor-Investigator, Gozdem Kayki, Investigator, Hacettepe University
Organization: Hacettepe University (Other)
Other Study IDs: go 20 334
Record Dates: First submitted 2020-09-03; First posted 2020-09-10 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: lung ultrasound — LUS was performed within first 20 to 30 minutes and repeated at 1, 2, 4 and 6 hours.

SUMMARY:
Lung ultrasonography (LUS) is fast and easy technique. it also has high reliability, so it has started to be used more in evaluating respiratory distress in the neonatal period. The most important feature of LUS is being radiation-free. Three LUS findings that show respiratory distress syndrome were described. They were white lung appearance, lack of preserved areas and loss of pleural integrity. The sensitivity of these findings was found to be 98-100% and the specificity 92-100%. A few studies have shown that surfactant need can be determined by LUS.

It was observed that lung findings were more severe in LUS performed in the early period because of non-completed fetal lung fluid clearence, but the findings could be improved during follow-up. Therefore, it is not known when the earliest time of LUS shows the actual clinical condition and course of the patient.

This study was planned to find the most reliable and earliest US time. Evaluation with LUS was done at 30 minutes and repeated at 1, 2, 4 and 6 hours of life. The LUS findings would be compared with x-ray findings and the correlation of surfactant need with LUS findings would also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* preterm babies with a gestational age 32 weeks or less
* babies treated with CPAP

Exclusion Criteria:

* If a baby was intubated in delivery room because of the responsiveness to face-mask ventilation, he/she was excluded.
* congenital heart diseases
* complex congenital malformations
* chromosomal abnormalities.

Ages: 30 Minutes to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: extreme preterm babies with a gestational age 32 weeks or less were admitted to NICU. Only babies who were treated with CPAP because of clinical signs of respiratory distress were enrolled the study.
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
lung ultrasound at 30 minutes | 30 minutes
  lung ultrasound findings
lung ultrasound at 1 hour | 1 hour
  lung ultrasound findings
lung ultrasound at 2 hour | 2 hour
  lung ultrasound findings
lung ultrasound at 4 hour | 4 hour
  lung ultrasound findings
lung ultrasound at 6 hour | 6 hour
  lung ultrasound findings

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kayki G, Yigit S, Tandircioglu UA, Celik HT, Yurdakok M. Lung ultrasound (LUS) and surfactant treatment: looking for the best predictive moment. J Perinatol. 2021 Jul;41(7):1669-1674. doi: 10.1038/s41372-021-01039-0. Epub 2021 Mar 23. PMID 33758395